CLINICAL TRIAL: NCT01595906
Title: The Affect of a Ventilated Helmet System on Human Physiological Load
Brief Title: The Affect of a Ventilated Helmet on Physiological Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1037-2011-IDF-CTIL
Record Dates: First submitted 2012-03-22; First posted 2012-05-10 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Physiological Strain
Keywords: Helmet; Heat Tolerance Test; ventilation System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The experiment subjects (Experimental): The subjects will undergo:
  1. 6 acclimatization days carried out by a standard protocol including a daily 2 hour effort performed in a climatic chamber, during which the subjects walk on a treadmill at 5km/h on a 2% incline under heat conditions (40 deg. centigrade & 40% RH). Core (rectal) and skin temperatures and heart rate will be monitored continuously.
  2. Three consecutive days including 3 scenarios:
     1. Without a helmet b.With a helmet c.With a ventilated helmet During the experiment days the subjects will be exposed to the following protocol : A 5 minute sitting, performing cognitive tests on a computer for 15 min, 120 min walking on a treadmill at 5km/h on a 2% incline, at the end of the effort the same cognitive tests will be repeated for extra 15 min, 155 min in total.
  Interventions: Procedure: Ventilated Helmet

INTERVENTIONS:
Procedure: Ventilated Helmet — The ventilation system is installed on the inner part of the helmet and connected to a bellows and an energy source placed on the vest worn by the soldier. The system's working principal is based on air perfusion with a small ventilator.

SUMMARY:
The use of infantry helmets under heavy heat stress conditions, during physical exertion, may hinder the body's ability to effectively dissipate heat from the head area, thereby damaging the soldier's function. Therefore head cooling may potentially enable a longer duration of activity until reaching fatigue. An improvement in function may also be possible.The purpose of this research is to determine the extent of the cognitive and physiological strain caused by wearing a helmet under exertional conditions while exposed to heavy heat stress and to evaluate the effect of a unique ventilation system connected to the helmet on strain reduction.

DETAILED DESCRIPTION:
12 young, healthy civilian volunteers, aged 21-28 will participate in the study. Following a day of examinations and 6 days of acclimatization in a climatic chamber in accordance with a well accepted protocol, the subjects will undergo 3 days of experiment that will include exposure to hot environmental conditions with different helmet-wearing scenarios, while wearing uniform and a combat vest: (a) without a helmet (b) with a helmet (c) with a helmet connected to a ventilation system. All 3 scenarios will include a two hour effort (walking on a treadmill) in heavy heat stress in the climatic chamber at our institute (the Heller institute of medical research).

ELIGIBILITY:
Inclusion Criteria:

* healthy civilian volunteers
* aged 21-28
* without known medical illnesses or medication use

Exclusion Criteria:

* the existence of or suspicion of existing cardiac or respiratory disease
* hypertension
* diabetes
* any hormonal disease or any other chronic illness that may inhibit participation in the experiment
* infectious disease 3 days prior to the experiment.

Ages: 21 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-10 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Physiological strain | 9 days
  The physiological strain will be determined by body core temperature and heart rate of the subjects during a heat tolerance test(HTT).

SECONDARY OUTCOMES:
Rectal temperature | 9 days
  The Rectal temperature will be mesured by a rectal thermistore during each HTT
Skin temperature | 9 days
  The Skin temperature will be mesured by skin thermistores on 4 sites (chest, leg and arm and head).
Heart Rate | 9 days
  Heart rate will be monitored using a polar watch.
Sweat Rate | 9 days
  Sweat rate will be calculated from the patient's weight and his water balance

CONTACTS AND LOCATIONS:
Overall Officials: Amit Druyan, M.D, Principal Investigator — IDF medical corps
Locations (1):
- Heller insitute, Sheba hospital, Ramat Gan, Israel